CLINICAL TRIAL: NCT02921243
Title: Schizophrenia and the Gut Microbiome
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Director, Maryland Psychiatric Research Cente, University of Maryland, Baltimore
Other Study IDs: HP-00069555
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metatranscriptomics: Metatranscriptomics analyses provide a snapshot of the expressed genes in a sample, which allows for mechanistic insights into the microbiome not possible with 16S rRNA profiling only.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stool Sample Collection
- Prebiotic

SUMMARY:
In a sample of 20 inpatients with a DSM-IV-TR/DSM 5 diagnosis of schizophrenia or schizoaffective disorder, investigators propose to conduct a prospective, 2 week observational trial to collect gastrointestinal stool samples in order to characterize the microbiota in people with schizophrenia and examine its variability over time. Participants may elect to participate for an additional two weeks, during which they will receive the prebiotic, oligofructose-enriched inulin (FOS), in order to examine its effects on the relative preponderance of butyrate-producing bacteria in the gut microbiome. Investigators will use an inpatient sample in order to standardize meals, exercise and environmental mediators. This is considered a feasibility, pilot study in order to apply for future grant funding. Investigators will recruit patients from the Treatment Research Program inpatient unit, Maryland Psychiatric Research Center, University of Maryland School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR /DSM 5 diagnosis of schizophrenia or schizoaffective disorder;
2. Age 18-64 years;
3. currently hospitalized for at least 7 days
4. currently treated with an antipsychotic, with no dose changes in last 14 days
5. ability to participate in the informed consent process, as determined by a score of 10 or greater on the Evaluation to Sign Consent

Exclusion Criteria:

1. Gastrointestinal disorders, including, but not limited to Crohn's Disease, Irritable Bowel Syndrome, Celiac Disease,
2. Organic brain disorder, including cerebrovascular accident; epilepsy; traumatic brain injury, Loss of consciousness (LOC) for more than 30 minutes
3. Mental retardation
4. Antibiotic or immune therapy within the last three months
5. Prebiotic or probiotic treatment within the last three months
6. Inability to understand English
7. Inability to cooperate with study procedures
8. Pregnant women
9. Prisoner status
10. For MRI ONLY Contraindication for MRI scanning (e.g. metal in body, pacemaker).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In-participants with Schizophrenia
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
16S rRNA gene amplicons from stool samples | 4 weeks
  The 16S rRNA gene amplicon data will be used to examine the relative preponderance of butyrate-producing bacteria in the gut microbiota of people with schizophrenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.mprc.umaryland.edu